CLINICAL TRIAL: NCT05884047
Title: The Effect Of Virtual Reality Glasses On Vital Signs And State Anxiety Level In Cancer Patients Receiving Chemotherapy For The First Time- Randomized Control Trial
Brief Title: The Effect Of Virtual Reality Glasses On Vital Signs And State Anxiety Level In Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahar İNKAYA (Other)
Responsible Party: Sponsor-Investigator, Bahar İNKAYA, Assoc. Prof., Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Ankara Yilidirim Beyazit Un.
Record Dates: First submitted 2022-01-21; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Cancer Patients
Keywords: Chemotherapy; Virtually Reality; Anxiety; Nursing
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Semi-experimental
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality glasses (Other): In the research, Samsung Gear VR SM-R323 brand and model SG glasses provided by the researcher were used. Patients were offered four different options to watch as "Forest of Serenity", "Calm Place", "Happy Place", "Gala 360 Travel & Relax". Forest of Serenity is a nature video consisting of bird sounds, colorful trees and flowers, and a clear lake where fish can be seen swimming in it. Calm Place is a relaxing video where cycles are shown 24 hours a day, where a person finds himself by the lake in the forest in snowy, rainy sunny weather. In Happy Place, one finds himself in a virtual camp environment where natural events such as dynamically changing weather, day-night cycles, and falling stars are experienced. Gala 360 Travel & Relax is a Paris-Notre Dame museum tour video.
  Interventions: Device: Virtual Glasses
- Scales (Other): Spielberger State Anxiety Inventory Vital Signs Follow-up Form
  Interventions: Device: Virtual Glasses

INTERVENTIONS:
Device: Virtual Glasses — In the research, Samsung Gear VR SM-R323 brand and model SG glasses provided by the researcher were used. Patients were offered four different options to watch as "Forest of Serenity", "Calm Place", "Happy Place", "Gala 360 Travel & Relax". Forest of Serenity is a nature video consisting of bird sounds, colorful trees and flowers, and a clear lake where fish can be seen swimming in it. Calm Place is a relaxing video where cycles are shown 24 hours a day, where a person finds himself by the lake in the forest in snowy, rainy sunny weather. In Happy Place, one finds himself in a virtual camp environment where natural events such as dynamically changing weather, day-night cycles, and falling stars are experienced. Gala 360 Travel & Relax is a Paris-Notre Dame museum tour video.

SUMMARY:
This study was conducted as a non-randomized control group experimental study to determine the effect of virtual reality glasses on vital signs and state anxiety levels.

DETAILED DESCRIPTION:
Purpose This study was conducted as a non-randomized control group experimental study to determine the effect of virtual reality glasses on vital signs and state anxiety levels in cancer patients receiving chemotherapy for the first time.

Methods and Sample The population of the study was composed of adult patients admitted to an oncology hospital in Ankara province with a diagnosis of stage I-II-III cancer to undergo chemotherapy treatment for the first time. The sample of the study consisted of 30 patients who were assigned to the intervention and control groups by the stratified sampling method (considering such characteristics as age, gender, marital status). The patient identification form, Spielberger state anxiety scale, patient opinion form, vital signs follow-up form, and virtual reality glasses were used to collect the data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stage 1,2,3 cancer
* Receive radiotherapy and chemotherapy for the first time
* Volunteer patients who agreed to participate

Exclusion Criteria:

-Patients outside the inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Vital signs- Blood pressure | first measurement just before the start of the chemotherapy infusion
  Systolic blood pressure values
Vital signs-pulse | first measurement just before the start of the chemotherapy infusion
  Pulse values
Vital signs- Blood pressure | the last measurement just after the end of the chemotherapy infusion
  Systolic blood pressure values
Vital signs-pulse | the last measurement just after the end of the chemotherapy infusion
  Pulse values

CONTACTS AND LOCATIONS:
Overall Officials: SEBILE OZDAG, Study Chair — Hacettepe University Adult Oncology Hospital
Locations (1):
- Bahar İnkaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No